CLINICAL TRIAL: NCT01568476
Title: Does Interneural Local Anesthetic Spread at the Site of Sciatic Nerve Bifurcation Shorten Block Onset Time?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 11-0059-A
Record Dates: First submitted 2012-03-06; First posted 2012-04-02 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Post Operative Analgesia; Regional Anesthesia; Sciatic Nerve Block
Keywords: Regional anesthesia; Sciatic nerve block; foot surgery; ankle surgery; Interneural local anesthetic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Distal (Active Comparator): Blockade of both terminal branches of Sciatic nerve separately, distal to bifurcation
  Interventions: Procedure: Distal
- Interneural (Active Comparator): sciatic nerve blockade at the site of bifurcation
  Interventions: Procedure: Interneural

INTERVENTIONS:
Procedure: Distal — Blockade of both terminal branches of Sciatic nerve separately, distal to bifurcation
  Arms: Distal
Procedure: Interneural — Sciatic nerve blockade at the site of bifurcation
  Arms: Interneural

SUMMARY:
Following foot and ankle surgery, ultrasound-guided sciatic nerve block (SNB) at the popliteal fossa decreases post-operative pain and opioid consumption. At the popliteal fossa, the sciatic nerve bifurcates to form the Common Peroneal Nerve (CPN) and Tibial Nerve (TN). Studies have shown that when both branches are blocked separately distal to the bifurcation site, block onset time is reduced by 30%. Through clinical observation, the investigators found that onset time is further shortened when ultrasound-guided SNB is performed at the site of bifurcation. This is because the local anesthetic spreads interneurally. The purpose of this study is to compare the block onset time of an ultrasound-guided sciatic nerve block at the site of nerve bifurcation with the blockade of each terminal nerve separately (TN and CPN) distal to sciatic nerve bifurcation.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* 18-85 years of age, inclusive
* 50-120 kg, inclusive
* 150 cm of height or greater

Exclusion Criteria:

* Contraindications to sciatic nerve block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the popliteal area)
* Significant peripheral neuropathy or neurological disorder affecting the lower extremity
* Pregnancy
* History of alcohol or drug dependency/abuse
* History of significant psychiatric conditions that may affect patient assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Block onset Time | every 5 minutes up to 45 minutes of the block or until surgery starts
  We aim to compare the block onset time of an ultrasound-guided sciatic nerve block at the site of nerve bifurcation resulting in interneural spread of local anesthetic with that of blockade of each terminal nerve separately (TN and CPN), distal to sciatic nerve bifurcation. We hypothesize that sciatic nerve blockade at the site of bifurcation with interneural local anesthetic spread within a common epineural sheath results in shorter onset time compared to blockade of each terminal nerve distal to sciatic nerve bifurcation.

SECONDARY OUTCOMES:
Extent of longitudinal local anesthetic solution spread | starting at block administration till 5 minutes after complete injection
Nerve diameter prior to and following injection | starting at block administration till 5 minutes after complete injection
Block procedure time | starting at block administration till complete injection(up to 10 minutes)
Number of skin punctures required. | starting at first attempt of block administration till complete injection(up to 10 minutes)
Block success rate | starting after complete injection up to 45 minutes
Incidence of block-related complications | immediately , at 24 hours and Post operative day 7
  Incidence of block-related complications (vascular puncture, hematoma formation, intravascular injection and post-operative neurologic deficit) will be documented, but due to the very low incidence in all block-related complications, this study is not powered to show a difference in safety
Postoperative pain | starting at patient's arrival at post-anesthetic care unit till 120 minutes
  Postoperative pain: Postoperative pain using a verbal rating score (0-10, where 0= no pain, 10=excruciating pain) at 0, 30, 60, 90 and 120 min upon admission to post-anesthetic care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada